CLINICAL TRIAL: NCT05063240
Title: Mobile Phone Text Messaging Plus Motivational Interviewing: Effects on Breastfeeding, Child Health and Survival Outcomes, a Group Sequential Randomised Standard of Care Controlled Trial
Brief Title: Mobile Phone Text Messaging Plus Motivational Interviewing: Effects on Breastfeeding, Child Health Outcomes
Acronym: MTM-MI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Stellenbosch (Other)
Collaborators: McMaster University (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Moleen Zunza, Dr, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: M21/03/010; TMA2020CDF-3169 (Other Grant/Funding Number: EDCTP2 supported by European Union and Fondation Botnar)
Record Dates: First submitted 2021-08-16; First posted 2021-10-01 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Breastfeeding, Exclusive; HIV Infections
Keywords: HIV; Infant feeding; mHealth; motivational interviewing; behavioural intervention
MeSH Terms: conditions — Breast Feeding; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile phone text messaging plus prospective motivational interviewing (Experimental): Experimental: Text messaging-motivational interviewing. Every Monday morning, a text message (SMS) will be sent to participants in the intervention group encouraging participants to continue breastfeeding, and inquire if participants have any problems breastfeeding the infants. Participants will be asked to respond within 48 hours, indicating no problem or a problem with breastfeeding that requires help. In addition to text messaging, participants will have motivational interviews post-delivery at weeks 2, 6, and 10. Motivational interviews will explore and support the participant's commitment to continue breastfeeding.
  Interventions: Behavioral: Mobile phone text messaging plus prospective motivational interviewing; Behavioral: Standard infant feeding counselling
- Standard infant feeding counselling (Active Comparator): Standard infant feeding counselling as part of routine primary healthcare practice
  Interventions: Behavioral: Standard infant feeding counselling

INTERVENTIONS:
Behavioral: Mobile phone text messaging plus prospective motivational interviewing — Interactive weekly mobile phone text messaging plus prospective motivational interviewing at study follow up visits
  Arms: Mobile phone text messaging plus prospective motivational interviewing
Behavioral: Standard infant feeding counselling — Standard infant feeding counselling as part of routine practice at primary healthcare facility

SUMMARY:
Background

Lack of breastfeeding, at a minimum, doubles the risk of infant death in the first six months of life. Many infants in low resourced settings at high risk of infectious disease morbidity and death are deprived of the immunological and nutritional benefits of breast milk, through an attenuated duration of breast milk exposure. South Africa has one of the lowest exclusive breastfeeding rates in Africa, 8% in infants under 6 months of age. Mobile phone text messaging as a simple, low-cost intervention improves medication adherence among patients with HIV, diabetes and tuberculosis. Motivational interviewing has been beneficial across many health problems, including HIV viral load suppression, body weight loss, and alcohol and tobacco use. Combining a number of intervention approaches is more likely to influence behaviour change than an individual approach. Investigators assume that continued breastfeeding is sustained among women living with HIV receiving weekly text messages combined with motivational interviewing and that this contributes to improved infant health outcomes.

Objectives:

1. To determine the effects of mobile phone text messaging combined with motivational interviewing versus standard of care on: (a) Continued exclusive breastfeeding to six month of child age, (b) Continued any form of breastfeeding to 6 month of child age.
2. To determine the contribution of the combined intervention on improved infant health outcomes: (a) Infant morbidity (all -cause hospitalization) and death (all -causes, (b) Infant growth.

Methods

Investigators propose a group sequential clinical trial to determine whether text messaging combined with motivational interviewing will prolong breastfeeding and the contribution of the combined intervention on improved infant health outcomes. The study will recruit 275 women living with HIV and HIV exposed infants at birth and randomly assign study interventions for 6 months.

DETAILED DESCRIPTION:
Background

In 2010, following changes to global HIV and infant feeding guidelines, the South African vertical transmission prevention program stopped provision of formula milk and adopted breastfeeding as the recommended infant feeding modality. However, in reality, there are short-falls in attaining optimal infant feeding practices, which are contributing to failure to achieving the Sustainable Development under-five child health targets in South Africa. It is essential for the well-being of women living with HIV and their infants to establish models for supporting optimal infant feeding practices to achieve the desired child health outcomes.

Despite several proven interventions to improve breastfeeding practices, in practice there is lack of progress in implementing these interventions to achieve optimal breastfeeding practices. Telephonic support and motivational interviewing have been beneficial across many health problems, including medication adherence among people living with HIV and to reduce alcohol and tobacco use. Investigators propose to combine telephonic support with motivational interviewing to support infant feeding among women living with HIV. Combining these two interventions has great potential; it is likely to be cost-effective, simple to implement and easily integrated within the established infant feeding counselling conventional models.

Objectives

1. To determine the effects of mobile phone text messaging plus motivational interviewing versus standard of care on: (a) Continued exclusive breastfeeding to six month of child age, (b) Continued any form of breastfeeding to 6 month of child age.
2. To determine the contribution of the combined intervention on improved infant health outcomes: (a) Infant morbidity (all -cause hospitalization) and all -cause death, (b) Infant growth.

Methods

Study design: Participants will be randomized in a 1:1 ratio using a permuted block method to receive study interventions versus standard of care for 24 weeks. Electronic sequence generation and random allocation will be done centrally. Participants meeting inclusion criteria who consent to participate will be enrolled and immediately assigned to a study arm sequentially.

Study interventions: All women and their infants, irrespective of study assignments, will receive health services and treatment according to the respective provincial guidelines applicable in the sector during the study. Participants will be evaluated soon after giving birth and post-delivery until cessation of breastfeeding or until end of the study.

Mobile phone text messaging: Every Monday morning, a research nurse will send text message to women in the intervention group encouraging mothers to exclusively breastfeed and inquire if mothers have any problems breastfeeding infants. Participants will be asked to respond by text within 48 hours, indicating no problem or a problem with breastfeeding and require help. The research nurse will review all the responses and then follow-up any participants who indicate a breastfeeding problem or call participants who fail to respond within 48 hours.

Motivational interviewing: In addition to text messaging, women will have individual motivational interviews post-delivery at weeks 2, 6, and 10. During the interviews, the research nurse will have to understand participant's frame of reference, reinforce participant's own self-motivational statements, monitor the readiness to change, and affirm the participant's freedom of choice. Advice will be given with participant's permission, and when given, the participant will make her own choice.

Usual standard of care: Participants randomized to the usual standard of care group will be counselled by primary healthcare nurses and trained lay counsellors to exclusively breastfeed for the first six months. Participants will be free to call the clinic staff at any time.

Sampling plan, recruitment, study assessment and follow-up: Pregnant women living with HIV and giving birth at a healthcare facility in Cape Town, South Africa, between October 2021 and September 2023 will be informed about the study and mothers who indicate interest in participating will be consented for the study. Informed consent will be requested to conduct an enrolment maternal interview, four in-person follow-up visits, child hospitalization medical record review, and child height and weight measurements.

Participants will have in-person follow-up at weeks 2, 6, 10, and 24 of child age. Research nurses or counselors will administer a baseline questionnaire and follow up study questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women living with HIV and HIV exposed infants
* initiating breastfeeding soon after delivery
* 18 years and older
* ownership of a mobile phone
* infant judged to be in good health who are discharged soon after delivery

Exclusion Criteria:

* initiating formula feeding soon after delivery
* multiple birth deliveries
* birthweight <2500
* gestational age <36 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who are exclusively breastfeeding | from birth to 6 month of child age
  Number of participants who report giving only breast milk and no other liquid or solid based foods to infants as assessed by the infant feeding questionnaire
Number of participants who are practicing any form of breastfeeding | from birth to 6 months of child age
  Number of participants who report giving breast milk and other liquid or solid based foods to infants as assessed by the infant feeding questionnaire

SECONDARY OUTCOMES:
Infant morbidity | from birth to 6 months of child age
  All -cause hospitalization and all -cause death
Infant weight in kilograms | from birth to 6 months of child age
  Infant weight measurements
Infant length in centimetres | from birth to 6 months of child age
  Infant length measurements

CONTACTS AND LOCATIONS:
Overall Officials: Moleen Dzikiti, Principal Investigator — University of Stellenbosch; Taryn Young, Study Chair — University of Stellenbosch; Mark Cotton, Study Chair — University of Stellenbosch; Lehana Thabane, Study Chair — McMaster University; Louise Kuhn, Study Chair — Columbia University
Locations (1):
- Khayelitsha District Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available on SUNScholarData, an institutional research data repository that is managed by Stellenbosch University library. Participant's anonymized and de-identified data will added to the public data repository.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available within 6 months of completing study follow up. Data will be available for 15 years.
Access Criteria: Researchers working on similar maternal-child health related studies with appropriate institutional review board approvals for any additional pooled analyses

REFERENCES:
- [Derived] Zunza M, Thabane L, Kuhn L, Els C, Lombard C, Cotton MF, Young T. A randomized controlled, trial on effects of mobile phone text messaging in combination with motivational interviewing versus standard infant feeding counselling on breastfeeding and child health outcomes, among women living with HIV. Int Breastfeed J. 2025 Jan 20;20(1):5. doi: 10.1186/s13006-024-00693-2. PMID 39833919
- [Derived] Zunza M, Thabane L, Kuhn L, Els C, Cotton MF, Young T. Mobile phone text messaging plus motivational interviewing versus usual care: study protocol for a randomized controlled trial to evaluate effects on breastfeeding, child health, and survival outcomes, among women living with HIV (MTI-MI). Trials. 2023 Oct 5;24(1):639. doi: 10.1186/s13063-023-07647-9. PMID 37794523